CLINICAL TRIAL: NCT06868654
Title: DREAMM 7: A Multicenter, Open-Label, Randomized Phase III Study to Evaluate the Efficacy and Safety of the Combination of Belantamab Mafodotin, Bortezomib, and Dexamethasone (B-Vd) Compared With the Combination of Daratumumab, Bortezomib and Dexamethasone (D-Vd) in Participants With Relapsed/Refractory Multiple Myeloma
Brief Title: China Subpopulation: Evaluation of Efficacy and Safety of Belantamab Mafodotin, Bortezomib and Dexamethasone Versus Daratumumab, Bortezomib and Dexamethasone in Participants With Relapsed/Refractory Multiple Myeloma
Acronym: DREAMM 7
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 207503-CHN
Record Dates: First submitted 2025-03-06; First posted 2025-03-11 (Actual); Results first posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-03

CONDITIONS: Multiple Myeloma
Keywords: China Subpopulation; Belantamab mafodotin; Relapsed/refractory multiple myeloma; Daratumumab; Bortezomib; Dexamethasone; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — belantamab mafodotin; daratumumab; Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Belantamab mafodotin and Bortezomib plus Dexamethasone (Experimental)
  Interventions: Drug: Belantamab mafodotin; Drug: Bortezomib; Drug: Dexamethasone
- Daratumumab and Bortezomib plus Dexamethasone (Active Comparator)
  Interventions: Drug: Daratumumab; Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Belantamab mafodotin — Humanized anti-B-cell maturation antigen (BCMA) antibody/drug conjugate
  Arms: Belantamab mafodotin and Bortezomib plus Dexamethasone
Drug: Daratumumab — Anti-cluster of differentiation 38 [CD-38] monoclonal antibody
  Arms: Daratumumab and Bortezomib plus Dexamethasone
Drug: Bortezomib — Proteasome Inhibitor
Drug: Dexamethasone — Synthetic glucocorticoid with anti-tumor activity

SUMMARY:
This study is designed to evaluate safety and efficacy of belantamab mafodotin in combination with bortezomib/dexamethasone versus daratumumab in combination with bortezomib/dexamethasone in the Chinese participants with relapsed/refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of multiple myeloma as defined by the International Myeloma Working Group (IMWG) criteria.
* Previously treated with at least 1 prior line of multiple myeloma (MM) therapy and must have documented disease progression during or after their most recent therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
* Must have at least 1 aspect of measurable disease, defined as one of the following;

  1. Urine M-protein excretion >=200 mg per 24-hour, or
  2. Serum M-protein concentration >=0.5 grams per deciliter (g/dL), or
  3. Serum free light chain (FLC) assay: involved FLC level >=10 mg per dL (>=100 mg per liter) and an abnormal serum free light chain ratio (<0.26 or >1.65).
* All prior treatment-related toxicities (defined by National Cancer Institute Common Toxicity Criteria for Adverse Events [NCI-CTCAE] version 5.0) must be <=Grade 1 at the time of enrollment, except for alopecia.
* Adequate organ function

Exclusion Criteria:

* Intolerant to daratumumab.
* Refractory to daratumumab or any other anti-CD38 therapy (defined as progressive disease during treatment with anti-CD38 therapy, or within 60 days of completing that treatment).
* Intolerant to bortezomib, or refractory to bortezomib (defined as progressive disease during treatment with a bortezomib-containing regimen of 1.3 mg/m^2 twice weekly, or within 60 days of completing that treatment). Note: participants with progressive disease during treatment with a weekly bortezomib regimen are allowed.
* Ongoing Grade 2 or higher peripheral neuropathy or neuropathic pain.
* Prior treatment with anti-B-cell maturation antigen (anti-BCMA) therapy.
* Prior allogenic stem cell transplant.
* Any serious and/or unstable pre-existing medical, psychiatric disorder or other conditions, including renal, liver, cardiovascular, or certain prior malignancies.
* Corneal epithelial disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2024-04-03 (Actual); Study Completion 2026-06-19 (Estimated)

CONTACTS AND LOCATIONS:
Locations (11):
- China (11):
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Changchun
  - GSK Investigational Site, Guangzhou
  - GSK Investigational Site, Hangzhou
  - GSK Investigational Site, Jinan
  - GSK Investigational Site, Nanjing
  - GSK Investigational Site, Shenyang
  - GSK Investigational Site, Suzhou
  - GSK Investigational Site, Tianjin
  - GSK Investigational Site, Wuhan
  - GSK Investigational Site, Zhengzhou

IPD SHARING:
Plan to Share IPD: No
GSK will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The results presented are until the primary completion date. Additional results will be provided within a year of study completion.
Groups:
- Belantamab Mafodotin + Bortezomib (Bor) + Dexamethasone (Dex): Chinese participants with Relapsed/Refractory Multiple Myeloma (RRMM) received intravenous (IV) infusion of 2.5 milligram (mg)/kilogram (kg) belantamab mafodotin on Day 1 of each 21-day Cycle until disease progression, intolerable toxicity, death, informed consent withdrawal, or study end, whichever comes first in combination with 1.3 mg/meter^2 (m^2) Bor administered subcutaneously (SC) once daily on Days 1, 4, 8 and 11 of each 21-day cycle along with 20 mg Dex via oral tablet or IV infusion once daily on Days 1, 2, 4, 5, 8, 9, 11, and 12 of each 21-day cycle for a total of 8 cycles.
- Daratumumab + Bor + Dex: Chinese participants with RRMM received 16 mg/kg Daratumumab IV infusion once weekly of each 21-day cycle in Cycle 1 to Cycle 3; once every 3 weeks on Day 1 of each 21-day cycle in Cycle 4 to Cycle 8; and once every 4 weeks on day 1 of each 28-day cycle from cycle 9 onwards until disease progression, intolerable toxicity, death, informed consent withdrawal, or study end, whichever comes first in combination with 1.3 mg/m^2 Bor administered SC once daily on Days 1, 4, 8 and 11 of each 21-day cycle along with 20 mg Dex oral tablet or IV infusion once daily on Days 1, 2, 4, 5, 8, 9, 11, and 12 of each 21-day cycle for a total of 8 cycles.
Period: Overall Study
Arm/Group | Belantamab Mafodotin + Bortezomib (Bor) + Dexamethasone (Dex) | Daratumumab + Bor + Dex
Started (Intent-to-Treat (ITT) Population included all randomized participants whether or not randomized treatment was administered.) | 32 | 40
Safety Population (Safety population included all randomized participants who took at least 1 dose of study treatment.) | 30 | 40
Completed | 0 | 0
Not Completed | 32 | 40
Not completed — Death | 4 | 14
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Physician Decision | 0 | 1
Not completed — Ongoing | 23 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Belantamab Mafodotin + Bortezomib (Bor) + Dexamethasone (Dex) | Daratumumab + Bor + Dex | Total
Number analyzed (Participants) | 32 | 40 | 72
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 63.0 (9.36) | 61.5 (8.95) | 62.2 (9.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 20 | 33
  Male | 19 | 20 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 32 | 40 | 72
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as time from randomization until earliest date of disease progression (PD), determined by Independent Review Committee (IRC), according to the International Myeloma Working Group (IMWG) Response Criteria, or death due to any cause. PD= increase of >=25% from lowest value in >=1 of following (serum M-protein [absolute increase >=0.5 grams per deciliter {g/dL}]; serum M-protein increase >=1g/dL [when lowest M-protein >=5g/dL]; urine M-protein [absolute increase >=200 milligrams per 24 hours {mg/24h}]; participants without measurable serum & urine M-protein levels, difference between involved & uninvolved serum free light chains (sFLC) levels [absolute increase >10mg/dL]; appearance of new lesion,>=50% increase from nadir in Sum of the products of the maximal perpendicular diameters of measured lesions (SPD) of >1 lesion, or >=50% increase in longest diameter of previous lesion >1 centimeter (cm) in short axis.
Time Frame: Up to approximately 32 months
Population: Intent-to-Treat (ITT) Population included all randomized participants whether or not randomized treatment was administered.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Belantamab Mafodotin + Bortezomib (Bor) + Dexamethasone (Dex) | Daratumumab + Bor + Dex
Number analyzed (Participants) | 32 | 40
Months | NA [20.2 to NA] — The median and upper limit 95% Confidence Interval were not estimable due to the length of follow-up in assessing the number of events. | 8.4 [4.9 to 21.5]
Statistical Analysis 1: Comparison: Belantamab Mafodotin + Bortezomib (Bor) + Dexamethasone (Dex) vs Daratumumab + Bor + Dex; Test type: Other; Hazard Ratio (HR) = 0.24, 95% CI 2-sided [0.11 to 0.56] — Hazard ratio was estimated using a Cox Proportional Hazards model stratified by the number of lines of prior therapy, prior bortezomib and revised international staging system (R-ISS) at screening, with a covariate of treatment

2. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as time from the date of randomization until the date of death due to any cause.
Time Frame: Up to 255 weeks
Reporting Status: Not Posted, anticipated posting 2027-06

3. Secondary Outcome: Duration of Response (DoR)
Description: DOR is defined as time from first documented evidence of partial response or better until first documented progression or death, whichever occurs first.
Time Frame: Up to 255 weeks
Reporting Status: Not Posted, anticipated posting 2027-06

4. Secondary Outcome: Minimal Residual Disease (MRD) Negativity Rate
Description: Minimal Residual Disease (MRD) negativity rate is defined as the percentage of participants who are MRD negative by next generation sequencing (NGS).
Time Frame: Up to 255 weeks
Reporting Status: Not Posted, anticipated posting 2027-06

5. Secondary Outcome: Complete Response Rate (CRR)
Description: CRR is defined as percentage of participants with a confirmed complete response (CR) or better (i.e., CR, stringent Complete Response (sCR)).
Time Frame: Up to 255 weeks
Reporting Status: Not Posted, anticipated posting 2027-06

6. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as percentage of participants with a confirmed partial response (PR) or better (i.e. PR, Very Good Partial Response [VGPR], CR or sCR).
Time Frame: Up to 255 weeks
Reporting Status: Not Posted, anticipated posting 2027-06

7. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: CBR is defined as percentage of participants with a confirmed minimal response (MR) or better per International Myeloma Working Group (IMWG).
Time Frame: Up to 255 weeks
Reporting Status: Not Posted, anticipated posting 2027-06

8. Secondary Outcome: Time to Response (TTR)
Description: TTR is defined as time from the date of randomization and the first documented evidence of response (PR or better) among participants who achieve partial response or better.
Time Frame: Up to 255 weeks
Reporting Status: Not Posted, anticipated posting 2027-06

9. Secondary Outcome: Time to Progression (TTP)
Description: TTP is defined as the time from the date of randomization until the earliest date of documented PD or death due to PD. PD= increase of >=25% from lowest value in >=1 of following (serum M-protein [absolute increase >=0.5 grams per deciliter {g/dL}]; serum M-protein increase >=1g/dL [when lowest M-protein >=5g/dL]; urine M-protein [absolute increase >=200 milligrams per 24 hours {mg/24h}]; participants without measurable serum & urine M-protein levels, difference between involved & uninvolved serum free light chains (sFLC) levels [absolute increase >10mg/dL]; appearance of new lesion,>=50% increase from nadir in Sum of the products of the maximal perpendicular diameters of measured lesions (SPD) of >1 lesion, or >=50% increase in longest diameter of previous lesion >1 centimeter (cm) in short axis.
Time Frame: Up to 255 weeks
Reporting Status: Not Posted, anticipated posting 2027-06

10. Secondary Outcome: Progression-free Survival on Subsequent Line of Therapy (PFS2)
Description: PFS2 is defined as time from randomization to disease progression after initiation of new anti-myeloma therapy or death from any cause, whichever is earlier. If disease progression after new anti-myeloma therapy cannot be measured, a PFS event is defined as the date of discontinuation of new anti-myeloma therapy, or death from any cause, whichever is earlier
Time Frame: Up to 255 weeks
Reporting Status: Not Posted, anticipated posting 2027-06

11. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA dictionary).
Time Frame: Up to 255 weeks
Reporting Status: Not Posted, anticipated posting 2027-06

12. Secondary Outcome: Number of Participants With Clinically Significant Changes in Hematology Parameters
Description: Blood samples will be collected for the analysis of hematology parameters.
Time Frame: Up to 255 weeks
Reporting Status: Not Posted, anticipated posting 2027-06

13. Secondary Outcome: Number of Participants With Clinically Significant Changes in Clinical Chemistry
Description: Blood samples will be collected for the analysis of clinical chemistry parameters.
Time Frame: Up to 255 weeks
Reporting Status: Not Posted, anticipated posting 2027-06

14. Secondary Outcome: Number of Participants With Clinically Significant Changes in Urine Dipstick
Description: Urine samples will be collected for the urine dipstick analysis.
Time Frame: Up to 255 weeks
Reporting Status: Not Posted, anticipated posting 2027-06

15. Secondary Outcome: Number of Participants With Abnormal Ocular Findings on Ophthalmic Examination
Time Frame: Up to 255 weeks
Reporting Status: Not Posted, anticipated posting 2027-06

16. Secondary Outcome: Plasma Concentrations of Belantamab Mafodotin (Total Antibody)
Description: Blood samples will be collected for PK analysis of belantamab mafodotin.
Time Frame: Up to 255 weeks
Reporting Status: Not Posted, anticipated posting 2027-06

17. Secondary Outcome: Plasma Concentrations of Belantamab Mafodotin (ADC)
Description: Blood samples will be collected for PK analysis of belantamab mafodotin.
Time Frame: Up to 255 weeks
Reporting Status: Not Posted, anticipated posting 2027-06

18. Secondary Outcome: Plasma Concentrations of Monomethyl Auristatin-F With a Cysteine Linker (Cys-mcMMAF)
Description: Blood samples will be collected for PK analysis of belantamab mafodotin.
Time Frame: Up to 255 weeks
Reporting Status: Not Posted, anticipated posting 2027-06

19. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibodies (ADAs) Against Belantamab Mafodotin
Description: Serum samples will be collected for the analysis of the presence of ADAs using validated immunoassays. All samples will be tested in screening assay, and positive samples will be further characterized for antibody titers.
Time Frame: Up to 255 weeks
Reporting Status: Not Posted, anticipated posting 2027-06

20. Secondary Outcome: Titers of ADAs Against Belantamab Mafodotin
Description: Serum samples will be collected for the analysis of the presence of ADAs using validated immunoassays. All samples will be further tested in screening assay, and positive samples will be further characterized for antibody titers.
Time Frame: Up to 255 weeks
Reporting Status: Not Posted, anticipated posting 2027-06

21. Secondary Outcome: Number of Participants With Maximum Post-baseline Change From Baseline in Individual Items of Patient-reported Outcome Version of the Common Term Criteria for Adverse Events (PRO-CTCAE)
Description: The PRO-CTCAE is a patient-reported outcome measure that was developed to evaluate symptomatic toxicities in patients in cancer clinical trials; it characterizes the frequency, severity, interference, and presence or absence of symptomatic toxicities. Responses can range from 0 ("never," "none," "not at all," or "absent") to 4 ("almost constantly," "very severe," or "very much"), with a higher score indicating a higher frequency, severity, or interference of adverse events.
Time Frame: Up to 255 weeks
Reporting Status: Not Posted, anticipated posting 2027-06

22. Secondary Outcome: Change From Baseline in Health Related Quality of Life (HRQoL) as Measured by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire 30-item Core Module (EORTC QLQ-C30)
Description: The EORTC QLQ-C30 includes 30-items with single and multi-item scales. These included five functional scales (physical functioning [PF], role functioning [RF], cognitive functioning [CF], emotional functioning [EF] and social functioning [SF]), three symptom scales (fatigue, pain and nausea/vomiting [N/V]), a global health status (GHS)/ Quality-of-Life (QoL) scale, and six single items (constipation, diarrhoea, insomnia, dyspnoea, appetite loss [AL] and financial difficulties [FD]). Response options are 1 to 4. Scores are averaged and transformed to 0 to 100, a high score for functional scales/ GHS/QoL represent better functioning ability or health-related quality-of-life (HRQoL), whereas a high score for symptom scales/ single items represent significant symptomatology. Baseline was defined as latest pre-dose assessment (Day 1) with a non-missing value, including unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Up to 255 weeks
Reporting Status: Not Posted, anticipated posting 2027-06

23. Secondary Outcome: Change From Baseline in HRQoL as Measured by EORTC IL52
Description: The EORTC Quality of Life Questionnaire 20-item Multiple Myeloma module (QLQMY20) is a supplement to the QLQ-C30 instrument used in participants with multiple myeloma. For the EORTC IL52, disease symptoms domain of the QLQ-MY20 will be used for bone aches or pain, back pain, hip pain, arm or shoulder pain, chest pain, and pain increasing with activity. The individual component scores in the disease symptom domain are averaged and transformed linearly to a score ranging from 0 to100. A high score for disease symptoms represents a high level of symptomatology or problems.
Time Frame: Up to 255 weeks
Reporting Status: Not Posted, anticipated posting 2027-06

ADVERSE EVENTS:
Time Frame: All cause mortality, non-serious adverse events (Non-SAEs) and serious adverse events (SAEs) were collected up to approximately 32 months. The results presented are until the primary completion date. Additional results will be provided within a year of study completion.
Description: Safety population included all randomized participants who took at least 1 dose of study treatment.
Arm/Group | Belantamab Mafodotin + Bortezomib (Bor) + Dexamethasone (Dex) | Daratumumab + Bor + Dex
All-Cause Mortality (participants affected / at risk) | 4/30 | 14/40
Serious Adverse Events (participants affected / at risk) | 25/30 | 27/40
Other Adverse Events (participants affected / at risk) | 30/30 | 39/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belantamab Mafodotin + Bortezomib (Bor) + Dexamethasone (Dex) (N=30) | Daratumumab + Bor + Dex (N=40)
Pneumonia (Infections and infestations) | 11 (17) | 6 (7)
Herpes zoster (Infections and infestations) | 2 (2) | 2 (2)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Febrile infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 9 (12) | 7 (8)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 7 (10) | 5 (5)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Reflux gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 3 (4) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Uveitis (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 2 (2) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngeal disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fracture pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypogammaglobulinaemia (Immune system disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vitrectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belantamab Mafodotin + Bortezomib (Bor) + Dexamethasone (Dex) (N=30) | Daratumumab + Bor + Dex (N=40)
Platelet count decreased (Investigations) | 23 (94) | 27 (79)
White blood cell count decreased (Investigations) | 16 (52) | 26 (93)
Alanine aminotransferase increased (Investigations) | 19 (45) | 19 (34)
Aspartate aminotransferase increased (Investigations) | 20 (79) | 15 (29)
Lymphocyte count decreased (Investigations) | 13 (57) | 22 (78)
Neutrophil count decreased (Investigations) | 14 (40) | 20 (58)
Gamma-glutamyltransferase increased (Investigations) | 12 (21) | 9 (17)
Blood lactate dehydrogenase increased (Investigations) | 11 (33) | 5 (15)
Weight decreased (Investigations) | 7 (9) | 7 (11)
Blood bilirubin increased (Investigations) | 5 (8) | 6 (16)
Blood creatinine increased (Investigations) | 4 (12) | 6 (19)
Blood alkaline phosphatase increased (Investigations) | 6 (13) | 2 (2)
Blood cholesterol increased (Investigations) | 2 (6) | 5 (23)
Blood pressure increased (Investigations) | 3 (5) | 2 (2)
Urine albumin/creatinine ratio increased (Investigations) | 4 (6) | 0 (0)
White blood cell count increased (Investigations) | 3 (4) | 1 (1)
Alpha hydroxybutyrate dehydrogenase increased (Investigations) | 3 (8) | 0 (0)
Bile acids increased (Investigations) | 3 (9) | 0 (0)
Blood urea increased (Investigations) | 3 (11) | 0 (0)
Electrocardiogram T wave abnormal (Investigations) | 2 (2) | 1 (1)
Neutrophil count increased (Investigations) | 2 (5) | 1 (1)
Blood bilirubin unconjugated increased (Investigations) | 0 (0) | 2 (5)
Blood glucose increased (Investigations) | 0 (0) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 20 (65) | 23 (84)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 13 (74) | 19 (104)
Hypocalcaemia (Metabolism and nutrition disorders) | 13 (32) | 16 (47)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 9 (30) | 14 (38)
Hyperglycaemia (Metabolism and nutrition disorders) | 6 (23) | 13 (28)
Hypophosphataemia (Metabolism and nutrition disorders) | 6 (12) | 13 (34)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 7 (12) | 10 (27)
Hyperuricaemia (Metabolism and nutrition disorders) | 8 (25) | 9 (33)
Hyponatraemia (Metabolism and nutrition disorders) | 6 (13) | 8 (13)
Hypermagnesaemia (Metabolism and nutrition disorders) | 3 (22) | 10 (49)
Decreased appetite (Metabolism and nutrition disorders) | 6 (8) | 6 (10)
Hypercalcaemia (Metabolism and nutrition disorders) | 4 (13) | 4 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 5 (18)
Hypoproteinaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (4)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (4) | 2 (2)
Hyperlipidaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 2 (13)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 19 (56) | 29 (72)
Thrombocytopenia (Blood and lymphatic system disorders) | 15 (63) | 13 (46)
Neutropenia (Blood and lymphatic system disorders) | 4 (9) | 4 (7)
Leukopenia (Blood and lymphatic system disorders) | 3 (7) | 2 (3)
Hypoglobulinaemia (Blood and lymphatic system disorders) | 2 (3) | 2 (4)
Lymphopenia (Blood and lymphatic system disorders) | 2 (12) | 2 (7)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 21 (29) | 14 (16)
COVID-19 (Infections and infestations) | 15 (19) | 14 (15)
Upper respiratory tract infection (Infections and infestations) | 11 (19) | 16 (24)
Herpes zoster (Infections and infestations) | 8 (10) | 3 (3)
Conjunctivitis (Infections and infestations) | 6 (11) | 2 (2)
Nasopharyngitis (Infections and infestations) | 5 (9) | 1 (1)
Bronchitis (Infections and infestations) | 1 (3) | 2 (2)
Skin infection (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (3) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 14 (24) | 13 (28)
Constipation (Gastrointestinal disorders) | 8 (11) | 10 (22)
Abdominal distension (Gastrointestinal disorders) | 6 (8) | 3 (7)
Flatulence (Gastrointestinal disorders) | 3 (3) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 4 (5) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 2 (2)
Toothache (Gastrointestinal disorders) | 3 (6) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Eructation (Gastrointestinal disorders) | 2 (8) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 7 (12) | 5 (5)
Malaise (General disorders) | 3 (3) | 8 (8)
Oedema peripheral (General disorders) | 5 (6) | 3 (5)
Asthenia (General disorders) | 3 (3) | 4 (4)
Fatigue (General disorders) | 2 (2) | 1 (1)
Vision blurred (Eye disorders) | 15 (44) | 1 (1)
Cataract (Eye disorders) | 8 (18) | 6 (7)
Foreign body sensation in eyes (Eye disorders) | 11 (37) | 0 (0)
Dry eye (Eye disorders) | 7 (25) | 2 (2)
Photophobia (Eye disorders) | 8 (20) | 0 (0)
Eye irritation (Eye disorders) | 5 (16) | 1 (1)
Visual acuity reduced (Eye disorders) | 5 (6) | 1 (1)
Lacrimation increased (Eye disorders) | 4 (7) | 1 (1)
Eye pain (Eye disorders) | 4 (21) | 0 (0)
Cataract cortical (Eye disorders) | 3 (3) | 0 (0)
Cataract nuclear (Eye disorders) | 1 (1) | 2 (2)
Visual impairment (Eye disorders) | 3 (5) | 0 (0)
Xerophthalmia (Eye disorders) | 3 (3) | 0 (0)
Eye discharge (Eye disorders) | 2 (2) | 0 (0)
Eye pruritus (Eye disorders) | 2 (6) | 0 (0)
Ocular hyperaemia (Eye disorders) | 2 (2) | 0 (0)
Pterygium (Eye disorders) | 0 (0) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 9 (9) | 10 (11)
Dizziness (Nervous system disorders) | 3 (3) | 3 (3)
Neuralgia (Nervous system disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 2 (3)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 18 (20)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 5 (6)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 8 (19) | 10 (14)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 5 (7) | 3 (3)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2024-10-17): https://cdn.clinicaltrials.gov/large-docs/54/NCT06868654/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-11): https://cdn.clinicaltrials.gov/large-docs/54/NCT06868654/SAP_001.pdf